CLINICAL TRIAL: NCT04765852
Title: Growth, Safety and Efficacy of a Probiotic Supplement: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Growth, Safety and Efficacy of a Probiotic Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20.11.INF
Record Dates: First submitted 2020-11-12; First posted 2021-02-23 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Probiotic Supplement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental): High dose probiotic supplement and maltodextrin as the excipient
  Interventions: Other: High dose probiotic supplement
- Experimental Group 2 (Experimental): Low dose probiotic supplement and maltodextrin as the excipient
  Interventions: Other: Low dose probiotic supplement
- Control Group (Placebo Comparator): Placebo supplement containing only maltodextrin but having the same appearance as the probiotic supplements
  Interventions: Other: Placebo

INTERVENTIONS:
Other: High dose probiotic supplement — One probiotic stick pack will be dissolved in 10 mL lukewarm formula milk or breastmilk at body temperature. The dissolved supplement will be fed orally, preferably in the morning, starting on Day 1 until Day 56.
  Arms: Experimental Group 1
Other: Low dose probiotic supplement — One probiotic stick pack will be dissolved in 10 mL lukewarm formula milk or breastmilk at body temperature. The dissolved supplement will be fed orally, preferably in the morning, starting on Day 1 until Day 56.
  Arms: Experimental Group 2
Other: Placebo — One placebo stick pack will be dissolved in 10 mL lukewarm formula milk or breastmilk at body temperature. The dissolved supplement will be fed orally, preferably in the morning, starting on Day 1 until Day 56.
  Arms: Control Group

SUMMARY:
The primary objective of the study is to demonstrate the safety of a daily high dose of a probiotic supplement by comparing the growth (weight gain, g/day) of formula-fed and/or breastfed infants in high dose group versus placebo group from enrolment to 8 weeks of intervention

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind study of healthy term infants, consisting of three randomized arms: placebo control group, high dose experimental group, and low dose experimental group. The study population, approximately 228, are infants 14 - 21 days of age who are formula-fed and/or breastfed who is aligned with the intended target population for a probiotic supplement. Placebo and probiotic supplements will be mixed with formula or breastmilk and fed orally using a feeding cup or syringe. All enrolled infants will participate in the trial for approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent document indicating that the infant's parent(s)/ legally accepted representatives LAR have been informed of all pertinent aspects of the study.
2. Infants whose parent(s)/LAR have reached the legal age of majority in the countries where the study is conducted.
3. Infants whose parent(s)/LAR are willing and able to comply with scheduled visits, and the requirements of the study protocol.
4. Infants whose parent(s)/LAR can be contacted directly by telephone throughout the study.
5. Infants whose parent(s)/LAR have access to a working freezer.
6. Infants must meet all the following inclusion criteria to be eligible for enrolment into the study:

   1. Healthy term (37-42 weeks of gestation) infant at birth.
   2. At enrolment visit, post-natal age 14-21 days (date of birth = day 0)
   3. Birth weight ≥ 2500g and ≤ 4500g.
   4. Breastfed and/or formula-fed infants (including exclusively and mixed fed breast- and formula-fed infants) whose parent(s)/LAR intent not to change the feeding regimen until the study end at 8 weeks of intervention.
   5. Formula-fed infants and their parent(s)/LAR must have independently elected, before enrolment not to breastfeed and their infant must tolerate a standard cow's milk infant formula not containing any probiotics at time of enrolment.

Exclusion Criteria:

1. Infants with conditions requiring specific infant feeding regimens other than those specified in the protocol.
2. Infants receiving complementary foods or liquids defined as 4 or more teaspoons per day or approximately 20 g per day of complementary foods or liquids at or prior to enrollment.
3. Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformations (e.g., cleft palate, extremity malformation).
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis).
   3. History of admission to the Neonatal Intensive Care Unit (NICU), except for admission for jaundice phototherapy.
   4. Other severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant inappropriate for entry into the study.
4. Infants who are presently receiving or have received prior to enrollment probiotic supplements or any of the following: medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool characteristics (e.g., glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g. insulin or growth hormone); gastric acid secretion.
5. Currently participating or having participated in another clinical trial since birth.

Ages: 14 Days to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Safety of high dose probiotic supplement (weight gain) | Day 56
  Compare the growth (weight gain, g/day) of formula-fed and/or breastfed infants in EG 1 vs. CG from enrolment to 8 weeks of intervention

SECONDARY OUTCOMES:
Efficacy of two different doses of probiotic supplement | Day 0, Day 25-27, Day 53-55
  Bifidobacteria abundance measured in the fecal sample collected at home after 8 weeks of intervention (V3) analyzed by next generation sequencing (NGS) technology.

OTHER OUTCOMES:
Additional growth parameters: weight | Day 0, Day 28, Day 56
  Weight in grams and corresponding weight-for-age Z-score according WHO growth standards
Additional growth parameters: length | Day 0, Day 28, Day 56
  Length in centimeters and corresponding length-for-age Z-score according WHO growth standards
Additional growth parameters: head circumference | Day 0, Day 28, Day 56
  Head circumference in centimeters and corresponding head circumference-for-age Z-score according WHO growth standards
Additional growth parameters: body mass index | Day 0, Day 28, Day 56
  BMI and corresponding BMI-for-age Z-score according WHO growth standards
Fecal microbiome composition | Day 0, Day 28, Day 56
  Overall fecal microbiota composition, diversity, and microbiota community types will be assessed using NGS technology (including relative abundance of beneficial bifidobacteria bacteria species and pathogenic bacteria species) and
Bifidobacteria colonization | Day 0, Day 28, Day 56
  Bifidobacteria colonization using a newly developed rapid diagnostic kit
Fecal microbiome: Continuation of bifidobacteria colonization | Day 84
  Continuation of bifidobacteria colonization 4 weeks after intervention stop using NGS technology and DNAFoil® technology
Fecal metabolic profile: Fecal pH | Day 0, Day 28, Day 56
  Fecal pH
Fecal metabolic profile: Fecal organic acids | Day 0, Day 28, Day 56
  Fecal organic acids (such as, but not restricted to lactate, propionate, butyrate, acetate, valerate, and total fecal organic acids)
Fecal metabolic profile: gut microbiota-derived metabolites | Day 0, Day 28, Day 56
  Concentration of gut microbiota-derived metabolites using mass spectrometry and/or nuclear magnetic resonance
Biological response of selected fecal metabolites | Day 0, Day 28, Day 56
  Biological response using cultured cell lines or combinations of cell lines (Cell-based functional assays)
Fecal markers of immune health and gut barrier | Day 0, Day 28, Day 56
  Total secretory IgA, calprotectin, and α-1-antitrypsin assessed by ELISA and Fecal cytokine levels (such as, but not restricted to: IL-1ra, IL-1α, IL-1β, IL-6, IFN- γ, and TNF-α) will be measured by multiplex assays
GI tolerance | Day 0, Day 28, Day 56
  Infant Gastrointestinal Symptom Questionnaire (IGSQ-13) Index Score for overall GI tolerance calculated from the IGSQ-13
GI-related behaviors: Stool frequency | Day 0, Day 25-27, Day 53-55
  GI endpoints will be recorded via the 1-day and 3-day GI Symptom and Behavior Diary
GI-related behaviors: Stool consistency | Day 0, Day 25-27, Day 53-55
  Stool consistency using a validated 5-point scale in the 1-day and 3-day GI Symptom and Behavior Diary
GI-related behaviors: Incidence of spitting-up | Day 0, Day 25-27, Day 53-55
  Incidence of spitting-up using a Likert scale via the 1-day and 3-day GI Symptom and Behavior Diary
GI-related behaviors: Incidence of flatulance | Day 0, Day 25-27, Day 53-55
  Flatulence of spitting-up using a Likert scale via the 1-day and 3-day GI Symptom and Behavior Diary
GI-related behaviors: Crying time | Day 0, Day 25-27, Day 53-55
  Crying time (hours/min) via the 1-day and 3-day GI Symptom and Behavior Diary
GI-related behaviors: Sleep time | Day 0, Day 25-27, Day 53-55
  Sleep time (hours/min) using a Likert scale via the 1-day and 3-day GI Symptom and Behavior Diary

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Foundation for Tropical Medicine, Inc., City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Undecided